CLINICAL TRIAL: NCT00237991
Title: A Multicentric, Post-Marketing Surveillance to Monitor the Safety and Reactogenicity of GlaxoSmithKline Biologicals Hepatitis A Vaccine Administered in Korean Population.
Brief Title: Safety of GlaxoSmithKline (GSK) Biologicals Hepatitis A Vaccine in Korean Population
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Other Study IDs: 104147
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Hepatitis A
MeSH Terms: conditions — Hepatitis A | interventions — Hepatitis A Vaccines

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Biological: Hepatitis A

SUMMARY:
GlaxoSmithKline Korea has submitted a registration file for its hepatitis A vaccine. The present study will collect clinical data in the local target population as per the requirement of Korean Food and Drugs administration (FDA).

DETAILED DESCRIPTION:
All subjects will be administered one dose of the hepatitis A vaccine.

ELIGIBILITY:
Inclusion criteria

* Subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol (e.g. be reachable over the phone) should be enrolled in the study.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Written informed consent is obtained from the subject/ subjects' parents or guardians.

Exclusion criteria

* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., Oral temperature < 37.5°C (99.5°F) / Axillary temperature < 37.5°C (99.5°F) / Rectal temperature < 38°C (100.4°F) / Tympanic temperature on oral setting < 37.5°C (99.5°F) / Tympanic temperature on rectal setting < 38°C (100.4°F).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline